CLINICAL TRIAL: NCT06046716
Title: A Preliminary Randomised Clinical Trial Looking at the Impact of State-mindful Self-compassion on Sexual Function Post-breast Cancer Treatments
Brief Title: The Impact of Mindful Compassion on Sexual Functioning Post Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Reader, London Metropolitan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LMU
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Sexual Functioning
Keywords: cancer; cancer treatment; wellbeing; sexual self efficacy; quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised control waitlist n=28 active experimental group and n=24 waitlist control delayed group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental mindful compassion group (Experimental): Experimental randomised controlled waitlist study The experimental group (n=28) will receive mindful compassion intervention at week 1 and intervention terminates at week 4
  Interventions: Behavioral: Mindful compassion based on behavioural change taxonomy experimental group
- Waitlist mindful compassion control group (Other): Experimental randomised controlled waitlist study The delayed group (n=24) will receive mindful compassion intervention at week 4 and intervention terminates at week 8
  Interventions: Behavioral: Mindful compassion based on behavioural change taxonomy experimental group

INTERVENTIONS:
Behavioral: Mindful compassion based on behavioural change taxonomy experimental group — Since this is a waitlist control study both groups get the same intervention. This is a mindful compassion intervention which is based on the behavioural change taxonomy techniques to support the reliability of the intervention. This will include sensate, mindful exercises, relaxation and attending to the critical voice. The intervention consists of behavioural, cognitive and mindful compassion constructs.

SUMMARY:
Sexual dysfunction is commonly reported post cancer treatments. Sexual desire and body image are interrelated. Indeed, sexual wellbeing can be affected by diagnosis, medication and cancer treatments which can damage body tissues such as the vagina or penis owing to radiation therapy, or insufficient lubrication caused by chemotherapy. Additionally, feeling sore, exhausted, anxious, depressed and 'not in the mood' further contribute to changes in sexual desire

Very few evidence-based online interventions have been developed to address sexual difficulties post cancer treatments. This extends to well-being, sexual self efficacy and quality of life. It is imperative that mindful compassion interventions are based on a behavioural taxonomy to support the reliability in the delivery of these interventions. Indeed, this study has set out to identify and describe the key components and behaviour change techniques as part of the online intervention. These have been mapped to a behaviour change taxonomy with the view of supporting standardisation for future trial implementation. Therefore, the aim of this study is to examine the effectiveness of an online mindful-compassion intervention using the 3-system model of emotions based on the behavioural taxonomy among a post cancer treatment group with the view of improving quality of life. The study intends to provide preliminary estimates of pre-post intervention on a waitlist controlled randomised controlled trial looking at sexual self-efficacy, well-being, sexual desire, mindfulness and self-compassion.

Quantitatively, the research is structured so that participants will be randomised to either the active experimental or delayed group. This intervention will be weekly for approximately 1 to 2 hours over 4 weeks. This A follow-up at 12 weeks will be taken to determine the sustainability of this intervention.

DETAILED DESCRIPTION:
Psychosocial interventions have varied in supporting post cancer treatments. An intervention gaining momentum in National Health Service practices is mindfulness. Mindfulness can mitigate negative self-thoughts and instead increase wellbeing and sexual self-efficacy which supports sexual functioning. Its applications are diverse and have extended to pre and post cancer treatment interventions. Benefits of mindfulness among post cancer treatment patients include lower levels of anxiety, depression and concerns regarding recurrence.

Mindful compassion is gaining popularity in health care. Mindful compassion consists of mindfulness, humanity, and self-kindness. Mindful compassion has been used in psychosexual services including varied sexual presentation such as sexual pain disorder. Indeed, the three systems model can be used to map out validate and normalise different emotional experiences - as well as map out how they can impact sexual arousal and enjoyment.

The intervention will be delivered by a qualified practitioner specialised in mindful compassion. Participants will be encouraged to engage with at home exercises including sensate, breathing exercises, sexual desire and fantasy diaries, mindfulness and self-compassion exercise including working with body image. This will be guided by the 3-system model of emotions where focus on mind and body will identify physiological changes to a perceived threat, to cognitively identify and attend to internal and external triggers and to incorporate mindful acceptance and compassion to address the critical inner voice. This will be applied to day to day living as well as applying this to sex, intimacy and body image. The foundation of the intervention will be based on a behavioural change taxonomy. This consists of 93 behaviour change techniques taxonomy in which the relevant taxonomies will be selected for this intervention. Table 1 outlines the foundation of the intervention. In total, 12 domains have been included in the development of this intervention. Of these, 20 out of the 93 Behaviour Change Techniques listed in the behaviour change techniques taxonomy were identified.

Table 1

Cognition

Psychosexual education - sex and cancer 1.1, 1.2, 1.3, 1.4 Understanding sexual well-being, efficacy, desire, fantasy and intimacy 1.1, 1.2, 1.3, 1.4, 4.1 Understanding mindful compassion- the threat and drive systems (inner critic) 4.1, 6.1, 7.1, 8.1, 8.7,11.2 Cognitive recognition of the internal and external triggers in relation to threat and drive 2.3, 7.1, 12.1, 13.2, 15.4 Recognition and reframe with acceptance (mind and body- soothing) 13.2, 13.4, 15.2, 15.4, 16.2 Mental rehearsal of fantasy, sensate or sex whether literal or imagery 11.2,15.2, 15.4, 16.2

Behavioural

Self-care Behaviours 3.3, 12.6, 13.1, 13.4 Self-monitoring towards goals 1.1, 1.3, 2.3 Graded tasks towards sensate, sexual fantasy or sexual practice 8.1, 8.7 Restructuring the physical environment (sex furniture, use of porn etc) 12.1 Breathing exercises to minimise distress and increase calmness and safety 8.1, 8.7, 16.2

Self-acceptance/compassion towards feeling soothed and nurtured

Valued self-identity (mind and body) 11.2, 13.1, 13.4 Using sensate to identify body change with acceptance 12.6, 13.1, 13.4 Understanding emotions, feelings and intimacy 3.3, 11.2, 13.1, 13.2, 13.4, 15.2, 15.4, 16.2 Self-directed meditation 4.1, 6.1,8.1, 11.2,15.2 Body scan - better awareness of mind and body (top to toe) 4.1, 6.1, 8.1, 11.2, 15.2 Mindfulness practices and being aware of the present moment 16.2 Mindfulness stretching focusing on mind and body connection 4.1, 6.1, 8.1, 11.2, 15.2 Self-compassion with positive self-identity and sexual embodiment post cancer treatments 11.2, 13.1, 13.2, 13.4, 13.5, 15.3, 15.4

Structuring of intervention (online once a week for 1 to 2 hours)

Week 0 (baseline measurements taken)

Week 1 Introduction - psychosexual education

Week 2 The three-model system of emotions and sexual functioning

Week 3 Sexual intimacy and the inner critic

Week 4 Embracing life and embodied sexuality post-cancer (commencement of the delayed group)

ELIGIBILITY:
Inclusion Criteria:

* Must be registered with a General Practitioner
* Must be registered with a healthcare service which supports post-cancer treatment
* Have sexual desire before cancer diagnosis
* Must be aged 18 years or older
* Must be able to read and write English
* Clinical diagnosis of cancer diagnosis via the National Health Service Services
* The Patient Health Questionnaire screening score would be between minimal to mild, 0-9.

Exclusion Criteria:

* Currently receiving cancer treatments
* Completed cancer treatments within six months
* Are not registered with a General Practitioner
* Are not registered with healthcare services providing post-cancer support
* Aged below 18 years old
* Reading and writing English difficulties
* Self-perceived low/minimal sexual desire before cancer diagnosis (lifelong)
* A terminal illness/end-of-life
* The Patient Health Questionnaire score range would be between moderate to severe, 10-27.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women participated in this study post breast cancer treatment
Enrollment: 52 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Patients Health Questionnaire | This is taken at week 0
  Measures levels of depression for inclusion and exclusion criteria. The score ranges between 0 and 27, with a higher score representing higher levels of depression.
Female Sexual Function Index | Weeks 0, 4 and 12
  This is a 19-item questionnaire on sexual function, including sexual desire, orgasm, lubrication, sexual satisfaction and pain. It has five response categories. Scores include severe 2-7.2, moderate 7.3-14.4, mild to moderate 14.5-21.6, mild 21.7- 28.1 cut-off value, and no female sexual dysfunction 28.2 -36.The lower the score, the higher the level of sexual dysfunction.
Adapted Sexual Self-efficacy Erectile Tool | Weeks 0, 4 and 12
  This is a 15-item questionnaire which focuses on sexual confidence and behaviour change associated with therapy. Participants' responses are measured by a 10-item scale ranging from 1 to 10 with 1 being the lowest level of self-efficacy and 10 is the highest. Scores range from 15 to 150 with higher levels representing higher levels of sexual self-efficacy. There is no reverse scoring.
The Short Warwick-Edinburgh Mental Wellbeing Scale | Weeks 0, 4 and 12
  A 7-item questionnaire with 5 response categories looking at functioning and feeling aspects of well-being. The response categories include 1=none of the time to 5=all of the time. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing.
The Brunnsviken Brief Quality of Life Scale | Weeks 0,4 and 12
  An 8-item questionnaire with five response categories looking at satisfaction with self, friends, family and creativity. The total score is calculated by summing the satisfaction ratings and summing the six products for a total score with score range between 0-96.
The Self-compassion Scale | Weeks 0, 4 and 12
  This is a 12-item measure with five response categories, 1 = almost never to 5= almost always, with higher scores indicating higher levels of self-compassion. The questionnaire measures self-kindness and self-judgement, common humanity and isolation, and mindfulness and over-identification with painful thoughts and emotions. Scores range between. An estimated score between 1-2.5 for overall self-compassion score indicates low levels of self-compassion. 2.5-3.5 indicates moderate. 3.5-5.0 means high levels of overall self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, PhD, Principal Investigator — London Metropolitan Univeristy
Locations (1):
- London Met university, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Result] Libman E, Rothenberg I, Fichten CS, Amsel R. The SSES-E: a measure of sexual self-efficacy in erectile functioning. J Sex Marital Ther. 1985 Winter;11(4):233-47. doi: 10.1080/00926238508405450. PMID 4078907
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Result] Spector IP, Carey MP, Steinberg L. The sexual desire inventory: development, factor structure, and evidence of reliability. J Sex Marital Ther. 1996 Fall;22(3):175-90. doi: 10.1080/00926239608414655. PMID 8880651
- [Result] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Result] Feldman, G., Hayes, A., Kumar, S., Greeson, J., & Laurenceau, J. P. (2007). Mindfulness and emotion regulation: The development and initial validation of the Cognitive and Affective Mindfulness ScaleRevised (CAMS-R). Journal of Psychopathology and Behavioral Assessment, 29(3), 177-190
- [Result] Neff, K. D. (2003). Development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250.
- [Result] Vosper, J., Irons, C., Mackenzie-White, K., Saunders, F., Lewis, R., & Gibson, S. (2021). Introducing compassion focused psychosexual therapy. Sexual and Relationship Therapy, 1-33.
- [Result] Saunders, F., Vosper, J., Gibson, S., Jamieson, R., Zelin, J., & Barter, J. (2022). Compassion Focused Psychosexual Therapy for Women Who Experience Pain during Sex. OBM Integrative and Complementary Medicine, 7(2), 1-1.
- [Result] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451